CLINICAL TRIAL: NCT02096757
Title: The Use of Fish Oil to Reduce Inflammation Caused by a Peripheral Vascular Intervention
Acronym: OMEGA-PVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-13123
Record Dates: First submitted 2014-03-22; First posted 2014-03-26 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Claudication; Critical Limb Ischemia; Endovascular procedure; Atherosclerosis
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Chronic Limb-Threatening Ischemia; Atherosclerosis | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Pro-Omega Placebo soybean capsules; 4.4gm/day (Nordic Naturals, Watsonville, CA, USA) 2 weeks prior to surgery and continued for 4 weeks after.
  Interventions: Other: Pro-Omega Placebo
- Pro-Omega (Experimental): High-dose, short-duration dietary omega-3 fatty acids supplementation; 325mg of EPA and 225mg of DHA per capsule. 4.4gm/day (Nordic Naturals, Watsonville, CA, USA) 2 weeks prior to surgery and continued for 4 weeks after.
  Interventions: Dietary Supplement: Pro-Omega

INTERVENTIONS:
Dietary Supplement: Pro-Omega — Pro-Omega (Nordic Naturals, Watsonville, CA, USA). Each ProOmega capsule contains 325mg of EPA and 225mg of DHA. 4.4gm/day 2 weeks prior to surgery and continued for 4 weeks after
  Other Names: Fish Oil
  Arms: Pro-Omega
Other: Pro-Omega Placebo — Placebo Comparator: soybean (Nordic Naturals, Watsonville, CA, USA); 4.4gm/day 2 weeks prior to surgery and continued for 4 weeks after
  Arms: Placebo

SUMMARY:
Investigators hypothesize that high-dose n-3 polyunsaturated fatty acids (PUFA) oral supplementation will improve will improve systemic inflammation and patency of peripheral vascular intervention (PVI).

DETAILED DESCRIPTION:
The OMEGA-PVI trial is a double-blind, randomized (2:1 active:placebo), placebo-controlled trial with 30 patients aged ≥ 40 years with PAD. Eligible patients will be screened according to specified inclusion and exclusion criteria. All patients will be treated per our current practice as reflected in the American Heart Association Practice guidelines on PAD. n-3 PUFA supplementation will be achieved with 4 capsules of Pro-Omega twice daily (Nordic Naturals, Watsonville, California, USA), corresponding to a total of 4.4g/day given prior to and immediately after the operation. Each ProOmega capsule contains 325mg of EPA and 225mg of DHA. The placebo group will take the same number of capsules containing inactive substance (soybean; Nordic Naturals), designed to be the same color and shape as the treatment capsules. Blood draws, questionnaires, and ultrasounds will be done periodically. Specific measurements will include established markers of inflammation and resolution of inflammation, as well as ultrasound measures of PVI patency. The study proposed here has the potential to provide important new insights on the role of nutritional interventions in PAD, as well as to improve outcomes related to surgical revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Disabling claudication or CLI as indication for PVI (Rutherford Class II-V)
* Objective evidence of PAD e.g. ABI < 0.9, TBI < 0.6 or absent pedal pulses
* Currently not taking high-dose n-3 PUFA, as defined by >2 g/day
* Able to provide written informed consent AND
* Undergoing a PVI (catheter-based therapy) involving the aorto-iliac segment, superficial femoral artery or popliteal artery.

Exclusion Criteria:

* Age < 40 or > 90 years
* Undergoing open surgical revascularization
* Evidence of active infection in limb or foot or osteomyelitis
* Extensive tissue loss (Rutherford Class VI Disease)
* Diagnosed hypercoagulable state
* Non-atherosclerotic/aneurysmal disease as indication for procedure
* Chronic liver disease or myopathy
* End-stage renal disease (CKD 5)
* Poorly controlled diabetes (HbA1C > 8%)
* Recent other major surgery or illness within 6 weeks
* Use of immunosuppressives or chronic inflammatory disorders
* History of organ transplantation
* Pregnancy or plans to become pregnant
* Condition in which patient life expectancy is less than one year

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Systemic Inflammatory bio-markers | 6 months
  Will reduce circulating pro-inflammatory markers (PIMs) and increase pro-resolution mediators (PRMs) assayed using targeted metabolo-lipidomics, increase PRM production within peripheral circulating monocytes.

SECONDARY OUTCOMES:
Safety | 6 months
  We hypothesize that n-3 PUFA supplementation in the peri-PVI period will be safe and will not lead to an increase in adverse events including bleeding and pseudoaneurysm formation.

OTHER OUTCOMES:
Primary patency | 6 months
  We hypothesize that n-3 PUFA supplementation in the peri-PVI period will lead to an improvement in the primary patency of PVI at 6 months, as demonstrated by ultrasound (U/S).

CONTACTS AND LOCATIONS:
Overall Officials: Warren Gasper, M.D, Principal Investigator — UCSF & SFVAMC
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Grenon SM, Hughes-Fulford M, Rapp J, Conte MS. Polyunsaturated fatty acids and peripheral artery disease. Vasc Med. 2012 Feb;17(1):51-63. doi: 10.1177/1358863X11429175. PMID 22363018
- [Background] Grenon SM, Aguado-Zuniga J, Hatton JP, Owens CD, Conte MS, Hughes-Fulford M. Effects of fatty acids on endothelial cells: inflammation and monocyte adhesion. J Surg Res. 2012 Sep;177(1):e35-43. doi: 10.1016/j.jss.2012.04.010. Epub 2012 Apr 27. PMID 22572621
- [Background] Grenon SM, Conte MS, Nosova E, Alley H, Chong K, Harris WS, Vittinghoff E, Owens CD. Association between n-3 polyunsaturated fatty acid content of red blood cells and inflammatory biomarkers in patients with peripheral artery disease. J Vasc Surg. 2013 Nov;58(5):1283-90. doi: 10.1016/j.jvs.2013.05.024. Epub 2013 Jul 2. PMID 23830313
- [Background] Grenon SM, Owens CD, Alley H, Chong K, Yen PK, Harris W, Hughes-Fulford M, Conte MS. n-3 Polyunsaturated fatty acids supplementation in peripheral artery disease: the OMEGA-PAD trial. Vasc Med. 2013 Oct;18(5):263-74. doi: 10.1177/1358863X13503695. Epub 2013 Sep 19. PMID 24052491
- See also: UCSF & SFVAMC Divisions of Vascular and Endovascular Surgery Clinical Trials — http://vascular.surgery.ucsf.edu/research/clinical-research/clinical-trials.aspx